CLINICAL TRIAL: NCT02958462
Title: Pre-myeloid Cancer and Bone Marrow Failure Clinic Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mrinal S. Patnaik, M.B.B.S., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16-004173; NCI-2022-07824 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Myeloid Malignancy; Inherited Bone Marrow Failure Syndrome; Clonal Expansion; Cytopenia; Bone Marrow Failure Syndrome; Clonal Cytopenia of Undetermined Significance; Clonal Hematopoiesis of Indeterminate Potential; Hematologic Neoplasms; Hematopoietic and Lymphatic System Neoplasm; Hereditary Neoplastic Syndrome; Idiopathic Cytopenia of Undetermined Significance; Idiopathic Dysplasia of Uncertain Significance; Low Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Congenital Bone Marrow Failure Syndromes; Cytopenia; Bone Marrow Failure Disorders; Hematologic Neoplasms; Neoplastic Syndromes, Hereditary | interventions — Specimen Handling; Biopsy; Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (biospecimen collection, NGS analysis) (Experimental): Participants may undergo blood sample collection, a bone marrow biopsy, a skin punch biopsy, hair follicle collection, a buccal swab, and/or saliva collection for NGS analysis on study. Patients may additionally undergo clinical assessment and may receive genetic counseling on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Punch Biopsy; Procedure: Buccal Swab; Other: Clinical Evaluation; Other: Genetic Counseling; Other: Quality-of-Life Assessment; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample, hair follicle, and saliva collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo a bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Punch Biopsy — Undergo a skin punch biopsy
  Other Names: BIOPSY, PUNCH; Punch Biopsy of Skin
Procedure: Buccal Swab — Undergo a saliva or buccal swab
  Other Names: Buccal Scraping; Buccal Smear; Buccal swab/scraping; Buccal Swabbing
Other: Clinical Evaluation — Undergo clinical assessment
  Other Names: Clinical Assessment
Other: Genetic Counseling — Receive genetic counseling
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment; QOL Assessment
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial tests next generation sequencing (NGS) for the detection of precursor features of pre-myeloid cancers and bone marrow failure syndromes. NGS is a procedure that looks at relevant cancer associated genes and what they do. Finding genetic markers for pre-malignant conditions may help identify patients who are at risk of pre-myeloid cancers and bone marrow failure syndromes and lead to earlier intervention.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To use genomics and functional translational studies to diagnose, prognosticate and potentially offer therapeutic directives for patients with precursor features of myeloid neoplasms (myelodysplastic syndrome [MDS], myeloproliferative neoplasms [MPN], MDS/MPN overlap syndrome) and germline predisposition/bone marrow failure states, who do not meet the criteria for the diagnosis of these cancers as of yet.

II. To identify patients with precursor myeloid malignancies and bone marrow failure syndromes.

III. To examine the utility of NGS methods for discovery of targets or pathways involved in precursor features of myeloid cancer and bone marrow failure.

IV. To use clinomics/genomics to better understand pathobiology and risk of disease progression.

V. To help better understand the implications of variants of unknown significance using computational biology and functional studies.

VI. To utilize normal, age and sex matched controls to validate genetic and epigenetic testing carried out under this protocol (essential for accurate data analysis).

VII. To assess frailty in patients with clonal hematopoiesis in order to validate genetic and epigenetic testing completed under this protocol as objective assessments of frailty and aging in comparison to standard of care frailty and geriatric assessments.

OUTLINE:

Participants may undergo blood sample collection, a bone marrow biopsy, a skin punch biopsy, hair follicle collection, a buccal swab, and/or saliva collection for NGS analysis on study. Patients may additionally undergo clinical assessment and may receive genetic counseling on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic cytopenias of unclear significance (ICUS)
* Patients with clonal hematopoiesis of indeterminate significance (clonal hematopoiesis of indeterminate potential [CHIP]), including the recently described CHIP syndrome called VEXAS (vacuoles, E1 ubiquitin ligase, X chromosomal, autoimmune and somatic)
* Patients with clonal cytopenias of undetermined significance (CCUS)
* Marrow failure syndromes with myeloid malignancy predisposition - telomere dysfunction, chromosomal breakage disorders
* Germ line inherited syndromes with risk for malignant transformation - GATA2, CEBPA, ETV-6, RUNX1, JAK2, PF6, etc.
* Low risk MDS (idiopathic dysplasia of unclear significance)
* Family member of a patient with one of the above conditions
* Patient at high risk or suspected of developing one of the above conditions

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-01-16 (Actual); Primary Completion 2030-09-15 (Estimated); Study Completion 2035-09-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of cytopenias | Up tof 5 years
  Assessed by the number of subjects whose cytopenias are persistent or progressive over the course of the study

SECONDARY OUTCOMES:
Occurrence of myelodysplastic syndrome (MDS) | Up to 5 years
  Assessed by the number of subjects who have evolved to MDS over the course of the study
Occurrence of acute myeloid leukemia (AML) | Up to 5 years
  Assessed by the number of subjects who have evolved to AML over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal S. Patnaik, MBBS, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials